CLINICAL TRIAL: NCT05189925
Title: NADPH Oxidase Correction in mRNA Transfected Granulocyte-enriched Cells in Chronic Granulomatous Disease (CGD)
Brief Title: NADPH Oxidase Correction in mRNA-transfected Granulocyte-enriched Cells in Chronic Granulomatous Disease (CGD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 220001; 22-I-0001
Record Dates: First submitted 2022-01-12; First posted 2022-01-13 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-10-16

CONDITIONS: Chronic Granulomatous Disease; Infection
Keywords: Primary Immune Deficiency; systemic infection; autologous transfusion; Apheresis
MeSH Terms: conditions — Granulomatous Disease, Chronic; Infections; Primary Immunodeficiency Diseases; Toxemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IV infusion of gp91-Grans at dose K: 1e6 cells/kg (Experimental): Adult CGD patients without systemic infection will participate in a dose-escalation trial to identify the most effective yet safe dose of study agent. Subjects enrolled will receive 1 administration of study agent at dose K, and safety of dose will be determined.
  Interventions: Biological: gp91 Grans
- IV infusion of gp91-Grans at dose K+1:1e7 cells/kg (Experimental): Adult CGD patients without systemic infection will participate in a dose-escalation trial to identify the most effective yet safe dose of study agent. Subjects enrolled will receive 1 administration of study agent at dose K+1, and safety of dose will be determined.
  Interventions: Biological: gp91 Grans
- IV infusion of gp91-Grans at dose K+2: 1-5e8 cells/kg (Experimental): Adult CGD patients without systemic infection will participate in a dose-escalation trial to identify the most effective yet safe dose of study agent. Subjects enrolled will receive 1 administration of study agent at dose K+2, and safety of dose will be determined.
  Interventions: Biological: gp91 Grans

INTERVENTIONS:
Biological: gp91 Grans — Adults with gp91phox-deficient CGD without systemic infection will participate in a dose escalation trial to identify the MTD (the most effective yet safe dose) of gp91 Grans IV infusion.

SUMMARY:
Background:

CGD is caused by a gene mutation. For people with CGD, their cells cannot kill germs well, so they can get frequent or life-threatening infections. Researchers want to see if a new procedure can help a person s cells kill germs for a short time. It uses messenger RNA (mRNA) to deliver correct instructions for the gene mutation to the cells.

Objective:

To test a procedure in which mRNA is added to a person s blood cells.

Eligibility:

Males aged 18-75 with CGD with a mutation in the gene that makes the protein gp91phox.

Design:

Participants will be screened with:

Medical history

Physical exam

Blood and urine tests

Swab to test for strep throat

Some screening tests will be repeated during the study.

Participants will be admitted to the NIH Clinical Center hospital for at least 7 days. They will have apheresis. For this, a medicine is injected under their skin to prepare their white blood cells for collection. An IV line is placed into an arm vein. Blood goes through the IV line into a machine that divides whole blood into red blood cells, plasma, and white blood cells. The white blood cells are removed, and the rest of the blood is returned to the participant through an IV line in their other arm. The next day, they will get their mRNA-corrected cells via IV. They will be monitored for 3 more days.

After discharge, participants will keep a symptom diary. They will be contacted weekly for one month, and then once a month. They will have a follow-up visit 3 months after the infusion.

DETAILED DESCRIPTION:
Study Design:

This is a phase 1, open-label, dose-escalation trial to assess the safety and feasibility of administering CGD-Grans to adult patients with X-linked CGD and to identify the maximum tolerated dose (MTD). Subjects will undergo granulocyte-enriched apheresis to provide cell product for mRNA-correction and then receive 1 administration of study agent. The first subjects enrolled will receive the study agent at the lowest dose, and when a level has been determined to be safe, the dose level will be increased to a second and then third dose level for subsequent subjects.Subjects will be hospitalized for at least 3 days after study agent administration and will return for a final study visit about 3 months after administration. Blood will be collected regularly for safety and research evaluations. The study hypothesis is that it is safe and feasible to administer mRNA-transfected autologous granulocyte-enriched apheresis product to restore protein expression and phagocyte nicotinamide adenine dinucleotide phosphate (NADPH) oxidase function in patients with CGD.

Study Agent Description:

The study agent is one administration of autologous CGD mRNA transfected granulocyte-enriched cells, referred to as CGD-Grans. The study agent is derived from apheresis product enriched for granulocytes, which are then transfected with CGD mRNA and administered as an intravenous (IV) infusion. CGD-Grans will be evaluated using the 3+3 modified Fibonacci model at the following 3 escalating dosages:

Dose K: 1 x 10^6 granulocyte-enriched cells/kg body mass

Dose K+1: 1 x 10^7 granulocyte-enriched cells/kg body mass

Dose K+2: 1-5 x 10^8 granulocyte-enriched cells/kg body mass

Each dose will be evaluated in at least 3 subjects. Dose escalation will be managed by a predetermined algorithm depending on the occurrence of drug-related toxicity (DRT). There will be at least 1 week between study agent administration to each subject.

Primary Objectives:

1. Determine the safety and feasibility of CGD-Grans infusion.
2. Determine an MTD for administration.

Secondary Objectives:

1. Assess efficacy of CGD-Grans at restoring NADPH oxidase.
2. Determine the kinetics of CGD-Grans.

Exploratory Objectives:

1. Assess for inflammatory responses to CGD-Grans infusion.
2. Assess for immune responses to protein expressed by the transfected mRNA.
3. Evaluate in vitro bactericidal activity of CGD-Grans.

Primary Endpoints:

1. Determine safety and feasibility by:

   Safety: Frequency of grade 3 or greater adverse events (AEs) or serious adverse events (SAEs) related to the study agent.

   Feasibility: Recruitment, implementation, and manufacturing of CGD-Grans for infusions.
2. MTD determination based on the rate of AEs. MTD is defined as the highest dose level that does not cause the same grade 3 or 4 AEs in 3 or more patients.

Secondary Endpoints:

1. Determine percent of circulating dihydrorhodamine (DHR) positive granulocytes following study agent infusion.
2. Serial measurement of circulating DHR+ granulocytes from peripheral blood until day 3 following study agent infusion or disappearance of DHR+ granulocytes.

Exploratory Endpoint:

1. Assess for increased expression of inflammation-related genes after study agent infusion.
2. Evaluate for development of antibodies against mRNA-expressed CGDphox.
3. Perform in vitro bactericidal activity of CGD-Grans.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals must meet all of the following criteria to be eligible for study participation:

* Males aged 18 to 75 years
* CGD confirmed by DHR and deficiency subtype confirmed by protein analysis and/or genetic sequencing
* Has a physician at home for follow-up care
* Able to provide informed consent
* For men who engage in activities that can result in pregnancy, agree to use contraception when engaging in sexual activities that can result in pregnancy. Contraception must be used from screening through 3 months after the CGD-Grans infusion. Acceptable methods of contraception include the following:

  * Hormonal contraception
  * Male or female condom

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

* Clinically unstable due to moderate to severe acute systemic infections as defined by persistent resting tachypnea, tachycardia, or hypoxia of >20% from baseline and hypotension.
* Current or history of stage 4 chronic kidney disease or estimated glomerular filtration rate [eGFR] <30 mL/min/1.73 m^2 within 90 days of baseline.
* Unstable diabetes mellitus with hemoglobin A1c >7.0% and fasting serum glucose >200 mg/dL at screening.
* Current or history of heart failure stage D as defined by the American College of Cardiology Foundation/American Heart Association guidelines.
* History of arrhythmias that are symptomatic and deemed clinically unsafe for participation by NIH CC Cardiology consultation.
* Current or history of invasive cancers that require chemotherapy within 5 years of screening.
* Active hepatitis B, C, or HIV infections at screening.
* Unstable hypertension requiring addition of new anti-hypertensives within 2 weeks of screening.
* Impaired renal function that is unstable, with serum creatinine >3.0 mg/dL and rising.
* Serum transaminases and bilirubin that are >3 x the upper limit of normal.

NOTE: For prospective subjects who, per PI assessment at screening, have abnormal liver function tests, and/or a significant history of liver disease, and/or liver-related complications of CGD, and who otherwise meet eligibility criteria [i.e. those who do NOT meet any of the exclusion set forth herein], a hepatology consult will be required at screening, and participation must be approved in writing by hepatology to the PI.

* Electrocardiogram abnormalities indicative of acute myocardial injury, or arrhythmias that presents anesthetic risks, at screening.
* Anemia with hemoglobin <8 g/dL (transfusions to correct anemia permitted).
* Thrombocytopenia (platelets <50 x10^9 cells/L) (platelet transfusions to correct thrombocytopenia permitted).
* Profound thrombocytopenia (platelet counts <10,000/microliter) that is not reversible with platelet transfusions.
* Abnormal prothrombin time/partial thromboplastin time (PT/PTT) values outside the ranges accepted at the NIH CC that are not corrected or that cannot be attributed to presence of Lupus anticoagulant (commonly found in CGD patients).
* Inherited bleeding disorder that precludes line placement.
* Severe oxygen-dependent pulmonary disease that increases risks of procedures that may require sedation.
* History of or current evidence of alcohol or illicit drug abuse or dependence.
* Participation in a clinical protocol that includes an intervention that, in the opinion of the investigator, may affect the results of the current study.

Subjects will be selected in an equitable manner from the available pool of potentially eligible individuals, without regard to factors such as gender, race, ethnicity, socioeconomic status, etc, except for age and sex.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Recruitment, implementation, and manufacturing of gp91-Grans for infusions. | 3 months
  Determine feasibility of gp91-Grans infusion.
MTD determination based on the rate of AEs. MTD is defined as the highest dose level that does not cause the same grade 3 or 4 AEs in 3 or more patients | 3 months
  Determine an MTD for administration.
Safety: Frequency of grade 3 or greater adverse events or serious adverse events related to the study agent | 3 months
  Determine safety of gp91-Grans infusion.

SECONDARY OUTCOMES:
Determine percent of circulating dihydrorhodamine (DHR) positive granulocytes following study agent infusion. | 3 months
  Assess efficacy of gp91-Grans at restoring NADPH oxidase
Serial measurement of circulating DHR+ granulocytes from peripheral blood until day 3 following study agent infusion or disappearance of DHR+ granulocytes. | 3 days
  Determine the kinetics of gp91-Grans.

CONTACTS AND LOCATIONS:
Overall Officials: Suk S De Ravin, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Marciano BE, Allen ES, Conry-Cantilena C, Kristosturyan E, Klein HG, Fleisher TA, Holland SM, Malech HL, Rosenzweig SD. Granulocyte transfusions in patients with chronic granulomatous disease and refractory infections: The NIH experience. J Allergy Clin Immunol. 2017 Aug;140(2):622-625. doi: 10.1016/j.jaci.2017.02.026. Epub 2017 Mar 22. PMID 28342916
- [Background] Stroncek DF, Leonard K, Eiber G, Malech HL, Gallin JI, Leitman SF. Alloimmunization after granulocyte transfusions. Transfusion. 1996 Nov-Dec;36(11-12):1009-15. doi: 10.1046/j.1537-2995.1996.36111297091747.x. PMID 8937413
- [Background] Heim KF, Fleisher TA, Stroncek DF, Holland SM, Gallin JI, Malech HL, Leitman SF. The relationship between alloimmunization and posttransfusion granulocyte survival: experience in a chronic granulomatous disease cohort. Transfusion. 2011 Jun;51(6):1154-62. doi: 10.1111/j.1537-2995.2010.02993.x. Epub 2010 Dec 22. PMID 21175646
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2022-I-0001.html